CLINICAL TRIAL: NCT01812460
Title: Progressive Resistance Training of the Extensor Muscle of the Thigh in COPD-patients Hospitalized With an Exacerbation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study had to stop due to organizational changes in Nordsjællands Hospital
Sponsor: Frederikssunds Hospital, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Frederikssunds Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-1-2012-085
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease; Muscle Atrophy
Keywords: COPD; muscle strength; resistance training; Physiotherapi; m. quadriceps; Acute exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention-training-group (Experimental): The patients begin training on day 1 of admittance. The training consists of knee extension performed in the sitting position on the bed with a 90 degrees of flexion of the knees. The weight cuffs are tired to the angles with a weight corresponding to 10 RM (the weight lifted 10 times) The weights and exercises are subjected to supervision on daily basis by the physiotherapist. The weight is increased after every session of training if more than 10 rep. can be performed with a given weight. Limitations to exercise is also recorded along with the degree of dyspnoe as assessed by the Borg CR10, possible oxygen supplementation and saturation is recorded before and following exercise.
  The weight cuffs are handed over to the patients for self guided exercise during weekends
  Interventions: Other: Intervention-training-group
- Control group (No Intervention): The patients randomized to the control group receive lung physiotherapy from day two of admittance. Lung physiotherapy consists of help to bring up sputum from the bronchi and lungs. The patients are instructed in breath exercises, use of Positiv Ekspiratory Pressure, breathing exercises, cough and pursed lip breathing. The patients are encouraged to spend as little time in bed as possible.

INTERVENTIONS:
Other: Intervention-training-group — As descriped in Arm Description
  Other Names: Training the knee ekstension with weight cuffs
  Arms: Intervention-training-group

SUMMARY:
We want to test the hypothesis, that resistance training by the use of weigth cuffs on the angle can prevent loss or improve the strength of the quadriceps muscle in COPD patients admitted to hospital due to an exacerbation. The training is started at day one of admittance and the strength of the quadriceps is measured by a portable dynamometer.

DETAILED DESCRIPTION:
Background Chronic obstructive pulmonary disease (COPD) is one of the most costly chronic diseases (1). In Denmark it can be estimated that approximately 400.000 people suffers from COPD amounting to about 15% of the adult population. COPD causes 10.000 visits to the emergency room, approx. 25.000 acute admissions to hospital and 3.500 deaths a year. The disease costs approx 2 billion Danish croners (400 million dollars) a year. Hospital admissions due to exacerbations adds to the most costly part of the disease burden to society. COPD is one of the few chronic diseases still on the rise (1).

COPD is characterized by an accelerated decline in lung function. Most of the patients with severe degree of COPD suffer from recurrent acute deterioration named exacerbations. An exacerbation is defined as a deterioration in symptoms including shortness of breath and sputum production leading to a chance in medical treatment. Frequent exacerbations are associated with an extra high rate of decline in lung function and a strongly negative impact on the quality of life. The disease progression is followed by a gradual loss in muscle mass and strength (3).

Admission to hospital has well known effects on maximal oxygen consumption and a reduction in the physical condition leads to a more severe degree of shortness of breath during physical activity (4). Just a few days in bed is followed by an important loss of muscle mass and strength. Immobilization causes a decrease in metabolism and a loss of active motor units and a reduced ability to activate the resting motor units. This has a greater negative impact on the strength in the extensors that are engaged in maintaining the upright position than other muscle groups. In keeping with this, the loss of muscle strength occurs at twice as high a rate in muscles of the lower limb than in those of the upper limb (5). This leads to an increased production of lactic acid and corresponding muscle fatique (6). Muscles engaged in knee extension loose strength at the highest rate during immobilization. This loss has great impact on the activities of daily life such as getting out of bed, rising from a chair and climbing stairs. Even though the patients regain their premorbide lung function and their symptoms improve to the "normal" level usually within 6 weeks, they do not reach their habitual level of physical activity as expressed by the 6MWT (7). Admittance due to exacerbations is followed by muscle wasting and prolonged inactivity, leading to an increased risk of recurrent exacerbations.

Physical training of the muscles is the most efficient treatment to maintain or increase muscle strength to prevent muscle wasting during immobilization. Since most of the decline in muscle strength occurs during the first days of bed rest - 3-4% per day - and most pronounced in the muscles of the lower limb, there is god reason for early intervention with physical training of the extensors of the lower limb, the earlier after admittance, the better.

There is solid evidence for a positive effect of training of clinically stable COPD patients. Only two studies have investigated the effect of training during admittance for an acute exacerbation (8) In the study by Troosters, the training consisted of 3 sets of 8 repetitions amounting to 70% of 1 repetition maximum (1RM: repetitions maximum: the maximal weight that can be handled only one time). The subjects had an FEV1 of 40 ± 12 % of predicted, and were trained by the use of a knee extension machine. We do not know the exact exclusion criteria of the study - did they include patients who were unable to move from the bed to the knee extension machine? Did the physiotherapists handled the most severely diseased patients differently? Moreover, it would be more general applicable, if the training could be performed with a less demanding and expensive equipment than a knee extension machine. Accordingly, there is a need for at study with a more detailed description of the training procedure, using a simple, low cost training device, that is applicable to many centers and hospital units.

Most patients suffering from a severe degree of COPD (GOLD III and IV) (3)will experience severe shortness of breath leading to exhaustion even after very low level activities. Unilateral resistance training of the quadriceps by the use of wrist weights is low cost, low technology.

The pilot study at our department of pulmonary medicine, Frederikssund Hospital, including 8 severely diseased COPD patients, trained by wrist weights on average for 5 days, showed that all patients improved their muscle strength - amounting to an average of 50%.

The study showed that progressive lower limb muscle exercise was possible even in the most severely disabled patients on home oxygen. We do not know if the surprisingly high degree of improvement should be ascribed to the training or other factors. Accordingly, we want to perform a randomized controlled single blinded study to clarify if progressive resistance training with wrist weights can improve the strength of the large extensor muscle of the lower limb to a degree that will translate into improved physical ability after discharge from hospital.

Randomizing The investigation is designed as a randomized, controlled, single blinded study. Patients who fulfill the inclusion criteria and none of the exclusion criteria are invited to participate in the study. After an initial evaluation and testing the patients are randomized to either standard pulmonary physiotherapy and physical training (intervention group) or standard physiotherapy without training (control group). The list of randomization is based on a computer program. Numbers of randomization are kept in 70 closed envelopes. The content of the envelope is disclosed only after inclusion, initial evaluation and testing. The envelopes are numbered on the outside (a consecutive line of numbers different from the numbers of randomization) and kept by a secretary and released in the order of outside number.

Tests at inclusion and after 6 weeks will be performed by physiotherapists blinded to the randomization. It is impossible to blind the physicians, nurses and physiotherapists at the pulmonary ward.

Security and Ethics Based on the current evidence, the patients are not exposed to any kind of risk, except that a slight degree of muscle soreness may occur following the first few days of physical training. The study is not blinded to the physiotherapists who perform the training, and if any problem related to training should occur, it will be easily addressed.

The present study aims at progressive physical training with cheap equipment which is easy to handle for both the physiotherapists and the patients with minimal risk to the patients. This adds to the importance of the study.

The control group will be treated according to usual therapeutic guidelines. The study is reported to the local ethical committee. The patients are covered by patient insurance of Frederikssund Hospital.

Registration of data and informed consent Data evaluation agrees to the technical demands made by the Danish Data Protection Agency The patients are familiar with all collected data, and information about this included in the informed consent.

All data of the study will be kept in a separate locked container in a locked room. Only the principal investigator has access to the room and container. Data will be stores in excel, where every patient has a unique number and all date from that particular patient is stored under this number. The security container is obtained for the specific purpose of the study and is in accordance with the procedures of the local region regarding login on the internet.

The patients will be contacted by the principal investigator or another member of the staff adequately trained for the study within 24 hours of admittance to the pulmonary ward of Frederikssund Hospital.

The patients will receive oral information and information in writing about the study the day of admittance, about their rights as voluntaries in a scientific study in the field of health science. The patient will be informed about the nature of the study according to the guidelines of The Danish Council of Ethics. The oral information is guided by the information in writing, where every aspect of the study is explained in detail to the patient. Informed consent is obtained the day after information after a minimum of 24 hours of reconsideration. The patient can decide to withdraw from the study at any time during the investigation. The investigators can also decide that a patient should be withdrawn from the study and the reason for exclusion should be documented in the research files.

Statistics The primary aim of the study is to compare the strength of the extensor of the thigh of the intervention group with that of the control group by an isometric contraction test.

Calculations have showed that the need for 35 subjects in each group to be able to reveal a difference in strength of at least 30%, with a limit of statistical significance of 5% and a power of 80%. The power calculation is based on the expected change in extension strength from the start of the study to discharge where it is not expected that the control group will improve in strength. .

The applied statistical analyses (by SPSS) will be repeated measures (ANOVA) to determine a systematic difference between muscle strenght with or without quadriceps training.

Measurements All participants are tested latest on day one after admittance, at discharge from hospital and on an outpatient basis 6 weeks later. The day of admittance is denoted as day 0. The 6 weeks follow up are chosen due to the belief that most COPD patients are clinically stable 6 weeks after an exacerbation.

Economy and Time schedule The study is started up by the persons responsible for the investigation. The study is not yet fully financed. We are planning to apply for additional finalcial support. None of the foundations will have any connection to the drug industry and none of the possible supporters will have any impact on the results, their interpretation or publication.

The study will start in autumn 2012 and finished when all 70 COPD patients are included and followed up, hopefully finished autumn 2013.

The results of the study both positive, negative and inconclusive will be reported in an international journal of pulmonary medicine. The results will be presented at relevant congresses both in Denmark and abroad

References

(1) Juel K, Døssing M. KOL i Danmark: sygdommen der hver dag koster 10 danskere livet. Kbh.: Statens Institut for Folkesundhed; 2003.

(3) GOLD- Guidelines. Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2011.. Available at: www.goldcopd.org. Accessed 26.06.12.

(4) Bernard S, LeBlanc P, Whittom F, Carrier G, Jobin J, Belleau R, et al. Peripheral muscle weakness in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med 1998 Aug;158(2):629-634.

(5) Bloomfield SA. Changes in musculoskeletal structure and function with prolonged bed rest. Med Sci Sports Exerc 1997 Feb;29(2):197-206.

(6) Steiner MC, Evans R, Deacon SJ, Singh SJ, Patel P, Fox J, et al. Adenine nucleotide loss in the skeletal muscles during exercise in chronic obstructive pulmonary disease. Thorax 2005 Nov;60(11):932-936.

(7) Pitta F, Troosters T, Probst VS, Spruit MA, Decramer M, Gosselink R. Physical activity and hospitalization for exacerbation of COPD. Chest 2006 Mar;129(3):536-544.

(8) Troosters T, Probst VS, Crul T, Pitta F, Gayan-Ramirez G, Decramer M, et al. Resistance training prevents deterioration in quadriceps muscle function during acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med 2010 May 15;181(10):1072-1077

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of COPD
* Be admitted to the pulmonary ward due to an exacerbation in COPD
* Provide informed consent to participation in the study
* Be able to maintain an upright position on a chair
* Be able to be guided to training and understand instructions for participating.

Exclusion Criteria:

* Patients suffering from diseases that prevents the use of wrist weights such as

  * Deep venous thrombosis (DVT)
  * Erysipelas
  * Painfull edema of the limbs And
  * Lack of ability to walk, habitually
  * Already participating in COPD rehabilitation program
  * Predicted hospital stay of less than tree days as predicted by a • pulmonary physician
  * Patients admitted Friday night or Saturday morning cannot be stared up within 24 hours of admittance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Maximal isometric knee extension power is measured unilaterally by a fixed dynamometer. | Dez. 2012 - dez. 2013
  To investigate if progressive resistance training with loose weights of the quadriceps muscle of COPD patients admitted due to an exacerbation will improve muscle strength more than a control group exposed to physiotherapy as usual i.e. without quadriceps training.

SECONDARY OUTCOMES:
3 functional test: Timed Up and GO(TUG), Sit to stand(STS) and 6 min.walk | dez 2012- dez 2013
  TUG: measures the time it takes to get up from the sitting position, walk 3 meter turn around, walk back and sit.
  STS: measures the number of times the patient can rise from a chair 43 cm to seat and sit during 30 seconds. The sit to stand test reflects the ability to deal with a very important part of every day life - to rise from a chair.
  6 min walk: how far can the patient walk in 6 min.

CONTACTS AND LOCATIONS:
Overall Officials: Linette M. Kofod, Phys.Ther, Principal Investigator — Frederikssund Hospital, Denmark; Martin Doessing, dr.med, Study Chair — Frederikssund Hospital, Denmark
Locations (1):
- Frederikssund Hospital, Frederikssund, Denmark